CLINICAL TRIAL: NCT06639880
Title: How Does Thoracic Spine Pathomechanics Disturb Lumbar Spine Mechanics? A Randomized Controlled Trial.
Brief Title: Thoracic Hyperkyphosis and Low Back Pain
Acronym: hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer of Biomechanics, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo University N
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: hyperkyphosis; Cobb's angle
MeSH Terms: conditions — Low Back Pain; Kyphosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): triple attack protocol which includes a modified P-A mobilization, manipulation, and stabilization program (Active and passive) for the thoracic spine in addition to the usual care and the core program for the lumbar spine
  Interventions: Other: triple attack protocol
- control (Active Comparator): the usual care for the lumbar spine which includes TENS, ultrasound, and myofascial release for the lumbar spine in addition to a core program including bridge, half bridge and clam shell exercise
  Interventions: Other: usual care exercise

INTERVENTIONS:
Other: usual care exercise — the usual care for the lumbar spine which includes TENS, ultrasound, and myofascial release for the lumbar spine in addition to a core program including bridge, half bridge and clam shell exercise
  Arms: control
Other: triple attack protocol — a modified P-A mobilization, manipulation, and stabilization program (Active and passive) for the thoracic spine in addition to the usual care and the core program for the lumbar spine
  Arms: study group

SUMMARY:
This study was conducted on forty male patients (15 in the control group and 25 in the study group)) with low back pain hyperkyphosis of the thoracic spine, ages ranged from 20 - 40 years old. The visual analogue scale, the Oswestry disability questionnaire, and Cobb's angle was assessed for all patients before any intervention and two months post-intervention.

DETAILED DESCRIPTION:
This study was conducted on 40 male patients aged 20 to 40 suffering from LBP. Patients were included in the study if they had hyperkyphosis with an X-ray cobb's angle greater than 40 degrees. The visual analogue scale (VAS), the Oswestry disability questionnaire (ODI), and Cobb's angle were assessed for all patients before and one month post-intervention. Patients who met the inclusion criteria and agreed to participate in this study were randomly assigned to one of the two groups. Group 1 (the control group) received the usual care for the lumbar spine which includes TENS, ultrasound, and myofascial release for the lumbar spine in addition to a core program including bridge, half bridge and clam shell exercise. Group 2 (the study group) received the triple attack protocol which includes a modified P-A mobilization, manipulation, and stabilization program (Active and passive) for the thoracic spine in addition to the usual care and the core program for the lumbar spine

ELIGIBILITY:
Inclusion Criteria:

* patients who has low back pain due to facet joint arthropathy or discogenic cause confirmrd by MRI. Chronic spine instability confirmed by clinical tests. Sacroiliac joint confirmed by claster of lattelets. Hyperkyphosis (>40 degree measured by cobb's angle)

Exclusion Criteria:

* any structural deformity (wedge fracture) or previous spinal surgeries. Spinal tumors or fracture or presence of active infection in the lumbar spine. Systematic disorder (Rheumatoid) Cauda equine lesion, the presence of any comorbidities such as hypertension, DM, hyperlipidemia, obesity, and any autoimmune disease, history of patients who suffered from cancer, unexplained weight loss, immunosuppression, prolonged use of steroids, intravenous drug use, urinary tract infection, pain that is increased or unrelieved by rest, fever, significant trauma related to age, bladder or bowel incontinence, urinary retention (with overflow incontinence), saddle anesthesia, loss of anal sphincter tone, major motor weakness in lower extremities, fever, and vertebral tenderness.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
level of percieved pain | six weeks
  The visual analogue scale used to evaluate level of percieved pain
thoracic kyphosis angle | six weeks
  x-ray cobb's angle used to evaluate the degree of hyper kyphosis of the lumbar spine

SECONDARY OUTCOMES:
degree of disability | six weeks
  the Oswestry disability questionnaire sued to evalute level of functional diability

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy, Giza
  - Faculty of physical Therapy Cairo University, Giza